CLINICAL TRIAL: NCT02800382
Title: Bronchoalveolar Lavage Liq To Distinguish Benign and Malignant Pulmonary Diseases
Brief Title: Paraoxanase Enzyme Activity in Patients With Pulmonary Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Mesut Subak, Chest Diseases Specialist Dr. Mesut Subak, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: Paraoxanaz
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Lung Diseases
Keywords: paraoxonase; lung diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung Malignancy (Other): Fiberoptic bronchoscopy was performed under local anaesthesia and sedation for taking Bronchoalveolar Lavage Liq for Paraoxanase activity. Blood samples were taken too.
  The samples (fine-needle aspiration biopsy and fine-needle aspiration cytology) were diagnosed by pathological examination.
  Interventions: Other: Take samples
- Lung bening Diseases (Other): Fiberoptic bronchoscopy was performed under local anaesthesia and sedation for taking Bronchoalveolar Lavage Liq for Paraoxanase activity. Blood samples were taken too.
  Interventions: Other: Take samples

INTERVENTIONS:
Other: Take samples — Fiberoptic bronchoscopy was performed under local anaesthesia and sedation for taking Bronchoalveolar Lavage Liq for Paraoxanase activity. Blood samples were taken too.

SUMMARY:
Lipid per oxidation final products and free oxygen radicals are thought as initiator role for developing of cancer in the body. Level of paraoxonase in the patients with cancer varies. In this research, the investigators investigated the contribution of level of serum and bronchoalveolar lavage paraoxonase in the differentiation of benign and malignant lung disease patients. This research includes the patients that are diagnosis of lung cancer (research group) and benign pulmonary disease (control group) participated by accepted fiberoptic bronchoscopy (FOB).

DETAILED DESCRIPTION:
Lipid per oxidation final products and free oxygen radicals are thought as initiator role for developing of cancer in the body. Level of paraoxonase in the patients with cancer varies. In this research, the investigators investigated the contribution of level of serum and bronchoalveolar lavage paraoxonase in the differentiation of benign and malignant lung disease patients. This research includes the patients that are diagnosis of lung cancer (research group) and benign pulmonary disease (control group) participated by accepted fiberoptic bronchoscopy (FOB).

Paraoxonase and Cancer Relations Oxidative stress is one of the important etiologic factor in carcinogenesis. Serum PON1 activity was found to be significantly lower in patients with lung cancer than healthy people by Elkiran and her friends et al. Also, gastroesophageal cancer, meningioma, high-grade glioma and ovarian epithelial was found to be significantly lower in tumour patients according to control groups in plasma. The relationship between serum PON1 level and the occurrence of cancer is still unknown. PON1 polymorphism has been reported to be related with an increased risk of occurrence of cancer in relation to environmental chemicals.

Reactive oxygen radicals can usually lead to tissue damage by attacking all cell components. Increased free oxygen radicals and oxidative stress which is formed in the body are one of the important risk factor in increasing various types of cancer. Lipid peroxidation's final products and scavenger system components are thought to have for a starter role in oncogenesis. Carcinogenic radicals that are liposoluble are formed as a result of lipid peroxidation and PON1 binds with radicals that are liposoluble. PON1 are thought to be capable to metabolize these radicals that are liposoluble. PON1 activity and oxidative stress has been suggested to be inversely related in serum and macrophages. Loss of paraoxonase protective effect may play a role in increasing the sensitivity to genomic damage which inflammatory oxidants and diets carcinogens caused .

Purpose of this research is to compare serum and bronchoalveolar lavage liqs PON contrasts between patients with lung cancer and the control group and to determine if the enzyme is lower in plasma and bronchoalveolar lavage liqs in case of malignant.

ELIGIBILITY:
Inclusion Criteria:

1. There are not any medical contraindications for fiberoptic bronchoscopy (FOB) and bronchoalveolar lavage(BAL)
2. Bronchoscopic symptom does not constitute an impediment status to performing.
3. The following method has been obtained in accordance with FOB and BAL material.

Exclusion Criteria:

1. The presence of a medical contraindication to FOB and BAL
2. During FOB not detecting or not technically making the suitable segment bronchus for BAL
3. Not to be duly provided BAL materials.

Inclusion criteria for the control(benign lung diseases) group;

1. Have lung disease without malignancy
2. The absence of addition disease
3. The absence of medical contraindications for FOB and BAL
4. The following method has been obtained in accordance with FOB and BAL material. Exclusion criteria for the control group;

1. Detection of a new addition disease or the presence of the addition disease 2. To have a medical contraindication to FOB or BAL 3. Not to be duly provided BAL materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Difference of Paraoxonase Serum and BAL Levels between malignant and benign lung diseases | 3 month
  Paraoxonase Measurement:
  Before bronchoscopy, 10 cc of blood were drawn from all patients via the cubital vein in sterile conditions. 16x100 mm Ayset tube was placed in two biochemistry tube. BAL material and a tube of blood sample were sent to The Microbiology Laboratory after the operation. The other one was sent to The Biochemistry Laboratory.
  Whole blood and BAL samples were centrifuged at 3500 rpm for 5 minutes in the laboratory and stocked at -200°C until the test run. Serum total cholesterol, HDL, LDL levels were researched at whole blood samples which are placed in another tube in biochemistry laboratory by using OLYMPUS AU 2700 autoanalyzer. For the measurement of PON levels in serum and BAL, Human Paraoxonase ELISA kit (Nova Tein Inc. Biosience. USA) was used.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Subak, MD, Study Chair — mesutsubak@gmail.com

IPD SHARING:
Plan to Share IPD: No
It can be shared, after being published in scientific journals.

REFERENCES:
- [Background] Gan KN, Smolen A, Eckerson HW, La Du BN. Purification of human serum paraoxonase/arylesterase. Evidence for one esterase catalyzing both activities. Drug Metab Dispos. 1991 Jan-Feb;19(1):100-6. PMID 1673382
- [Background] MAZUR A. An enzyme in animal tissues capable of hydrolysing the phosphorus-fluorine bond of alkyl fluorophosphates. J Biol Chem. 1946 Jul;164:271-89. No abstract available. PMID 20989488
- [Background] Geldmacher-von Mallinckrodt M, Diepgen TL, Duhme C, Hommel G. A study of the polymorphism and ethnic distribution differences of human serum paraoxonase. Am J Phys Anthropol. 1983 Nov;62(3):235-41. doi: 10.1002/ajpa.1330620302. PMID 6318563
- [Background] Humbert R, Adler DA, Disteche CM, Hassett C, Omiecinski CJ, Furlong CE. The molecular basis of the human serum paraoxonase activity polymorphism. Nat Genet. 1993 Jan;3(1):73-6. doi: 10.1038/ng0193-73. PMID 8098250
- [Background] Mackness B, Durrington PN, Mackness MI. Human serum paraoxonase. Gen Pharmacol. 1998 Sep;31(3):329-36. doi: 10.1016/s0306-3623(98)00028-7. PMID 9703197
- [Background] Krzystek-Korpacka M, Boehm D, Matusiewicz M, Diakowska D, Grabowski K, Gamian A. Paraoxonase 1 (PON1) status in gastroesophageal malignancies and associated paraneoplastic syndromes - connection with inflammation. Clin Biochem. 2008 Jul;41(10-11):804-11. doi: 10.1016/j.clinbiochem.2008.03.012. Epub 2008 Apr 4. PMID 18423402
- [Background] Griffin PE, Roddam LF, Belessis YC, Strachan R, Beggs S, Jaffe A, Cooley MA. Expression of PPARgamma and paraoxonase 2 correlated with Pseudomonas aeruginosa infection in cystic fibrosis. PLoS One. 2012;7(7):e42241. doi: 10.1371/journal.pone.0042241. Epub 2012 Jul 31. PMID 22860094